CLINICAL TRIAL: NCT02559934
Title: An Open-label, Multiple-dose, Pharmacokinetic Study of SR-T100 Gel (Containing 2.3% Solamargine in Solanum Undatum Plant Extract) in Patients With Actinic Keratosis
Brief Title: Multiple-dose Pharmacokinetic Study of Solamargine in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GESRTAKD
Record Dates: First submitted 2015-08-11; First posted 2015-09-25 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — beta-solamarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SR-T100 gel (Experimental): A single dose of 0.3-0.5 g topical SR-T100 gel (containing 2.3% solamargine in Solanum undatum plant extract) in 25 cm2 skin area covered by an occlusive dressing at least 20 hours a day and will be given once daily for sixteen consecutive weeks.
  Interventions: Drug: SR-T100 Gel

INTERVENTIONS:
Drug: SR-T100 Gel — 0.3-0.5 g topical SR-T100 gel (containing 2.3% solamargine in Solanum undatum plant extract)
  Other Names: Solamargine

SUMMARY:
The aim of this study is to assess the delivery of SR-T100 from the topical gel (containing 2.3% solamargine in Solanum undatum plant extract) by determining the plasma levels of solamargine in subjects with AK while administration of a 25 cm2 contiguous or non-contiguous dermal treatment area.

DETAILED DESCRIPTION:
It is an open-label, multiple-dose, pharmacokinetic study. In stage 1, plasma concentration of solamargine will be examined after the test products were administrated to 5 subjects with Actinic Keratosis (AK). Thereafter, an interim report based on the results of stage 1 will be submitted for Taiwan Center for Drug Evaluation (CDE) review to determine stage 2 will be conducted or not. For stage 2, another 5 subjects with AK will be enrolled to complete the study.

The subjects will be recruited from AK patients of Taiwan. All subjects will sign an informed consent form (ICF). A copy of the signed ICF will be handed to the subjects. The subjects will be screened on an outpatient basis within 1 month prior to entry according to defined inclusion and exclusion criteria (medical history, personal history, physical examination, and laboratory values). The subject must be qualified for the study by fulfilling all of the inclusion and none of the exclusion criteria.

In the study period, study drug will be given once daily for sixteen consecutive weeks. Specifically, subjects will receive a single dose of 0.3-0.5 g topical SR-T100 gel (containing 2.3% solamargine in Solanum undatum plant extract) in 25 cm2 skin area covered by occlusive dressing at least 20 hours a day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female is 20 years of age or above.
* Patient has AK lesions located within a 25 cm2 contiguous or non-contiguous treatment area.
* Patient has at least one clinical confirmed AK lesion within the selected treatment area before.

Exclusion Criteria:

* Patient had used the following treatments within 4 weeks prior to the study treatment initiation: immunomodulators or immunosuppressive therapy, interferon or cytotoxic drugs.
* Patient had treated with topical 5-FU, diclofenac gel, imiquimod, ingenol mebutate, corticosteroids, retinoids or masoprocol on the treatment area within 4 weeks prior to the study treatment initiation.
* Patient had received cryodestruction, chemodestruction, curettage, photodynamic therapy or surgical excision on the treatment area within 4 weeks prior to the study treatment initiation.
* Patient had received any of the following treatments on the treatment area in the 6 months before study treatment initiation: psoralen plus Ultraviolet A therapy, Ultraviolet B therapy, laser abrasion, dermabrasion, chemical peel.
* Patient had used any topical preparations, such as sunscreens, moisturizers, body oils, or alpha or beta hydroxyl acids, in the treatment area within 24 hours before and during the study course.
* Patient is known to be hypersensitive to the study medication.
* Female who is pregnant, breast-feeding or considering becoming pregnant while during the study.
* Donation of 500 ml of blood in the past 3 months prior to dosing or donation of 250 ml of blood in the past 2 months prior to dosing.
* Patient had used of any investigational drug within the past 30 days before enrollment.
* Patient has any dermatological disease and/or condition, such as atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, melanoma, or other possible confounding skin conditions in the treatment or surrounding area (5 cm distances from treatment area).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2019-01 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
AUC0-τ,ss; | sixteen consecutive weeks.
  AUC0-τ,ss was determined by the area under the plasma concentration-time curve during a dosing interval at the last dose determined by the trapezoidal rule
AUMC0-τ,ss | sixteen consecutive weeks.
  AUMC0-τ,ss was determined by the area under the plasma (first) moment concentration-time curve during a dosing interval at the last dose determined by the trapezoidal rule according to the following equation:
  AUMC0-τ,ss = Σ[(tn - tn-1)(Cn-1tn-1 + Cntn) /2]
Cmax,ss; | sixteen consecutive weeks.
  Cmax,ss was determined by the the highest observed plasma concentration at steady state (the last dosing interval)
Cmin,ss; | sixteen consecutive weeks.
  Cmin,ss was determined by the minimum observed plasma concentration at steady state
Cave,ss | sixteen consecutive weeks.
  Cave,ss was determined by the average plasma concentration at steady state (the last dosing interval) according to the following equation:
  Cave,ss = AUCss / dosing interval
Fluctuation | sixteen consecutive weeks.
  Fluctuation was determined by the Fluctuation index of concentration at steady state
Tmax,ss; | sixteen consecutive weeks.
  Tmax,ss was determined by the time to reach highest observed plasma concentration at steady state (the last dosing interval)
kel | sixteen consecutive weeks.
  kel was determined by the plasma elimination rate constant determined by simple linear regression based on the terminal phase of plasma concentration
T½; | sixteen consecutive weeks.
  T½ was determined by the plasma half-life estimated by (0.693/kel)
MRTss | sixteen consecutive weeks.
  MRTss was determined by the mean residence time determined by AUMC0-τ,ss / AUC0-τ,ss

SECONDARY OUTCOMES:
Adverse events will be recorded to evaluate the safety outcome. | sixteen consecutive weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kou-Wha Kuo, PhD, Study Director — G&E Herbal Biotechnology Co., LTD
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan